CLINICAL TRIAL: NCT04511949
Title: Epidemiological Study of the Spread of SARS-CoV-2 in the Household of a Person Who Has Had a COVID-19 Disease
Brief Title: COVID-19: Epidemiological Study of the Spread of SARS-CoV-2 in the Household of a Person Who Has Had a COVID-19 Disease
Acronym: FAMICOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CREPATS 012
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional, single-center study carried out on the cohort of index patients followed on an outpatient basis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No arm (Other): No arm
  Interventions: Diagnostic Test: COVID-19 IgG / IgM rapid test (whole blood, serum, plasma)

INTERVENTIONS:
Diagnostic Test: COVID-19 IgG / IgM rapid test (whole blood, serum, plasma) — * The rapid test is performed using a drop of blood obtained at the fingertip (10 microliters) using a lancet.
  * The dropper pipette, held vertically, collects the drop of whole blood up to the "sample line"
  * Place 1 drop of whole blood (10 μL in the sample well (S) of the cassette.
  * Immediately add 2 drops (80μL) of buffer to the well (B) of the cassette.
  * Avoid air bubbles; if there is an air bubble, add a 3rd drop of buffer.
  The reading is taken after 10 minutes at most by the healthcare professional under medical supervision.
  In case of sepositivity of the rapid test, it may be offered to index cases and adult contacts, a blood sample of 5 ml of blood for a serothèque allowing a characterization of the antibodies and in particular of the neutralizing antibodies.

SUMMARY:
Evaluating the rate of exposure to the virus in the close contact population who shared the home of a person infected with SARS-CoV-2 at the time of infection of the index case - adults or children - is a major factor in assessing the spread. virus in the family environment, assess the factors of circulation and determine whether immunity has been acquired. Screening for specific antibodies to SARS-CoV-2 will determine the exposure and protection acquired against this virus.

Knowing the intra-family secondary transmission rate is essential for supporting the strategies for lifting the confinement envisaged and implementing a personalized approach.

As of March 8, a platform for the home management of COVID + patients was set up when they, pauci or moderately symptomatic, do not require hospitalization. As of May 6, 2020, 881 patients have been registered in COVID and followed, constituting the active COVIDOM / PSL file. Of the 512 patients included between March 1 and 31, 45% have a household consisting of 3 people.

All patients had weekly clinical follow-up by telephone for the duration of the disease with a maximum of 4 weeks having been achieved.

If the recommendations of barrier gestures, isolation in an apartment were made during the symptomatic phase, the absence of masks available to all did not allow, in practice, to achieve the isolation and quarantine recommended ideally. to break the transmission of the virus.

The FAMI-CoV study proposes to assess the rate of exposure to the virus in contacts sharing the same focus of index cases. A sub-study will assess the proportion of antibodies that have been neutralizing.

DETAILED DESCRIPTION:
Transmission of the virus is possible from patients without or with very few symptoms. The viral load is high from the onset of symptoms and then decreases to the limit of detection on D21. The period of contagiousness would start 2.3 days before the symptoms (95% CI, 0.8-3.0 J) and would reach a peak at 0.7 J (95% CI, -0.2-2.0 J). This contagiousness would then decrease rapidly within 7 days with an estimated proportion of pre-symptomatic transmission of 44%.

The IgG and IgM antibodies generated by SARS-CoV-2 can be detected 1 to 3 weeks after exposure.

Guo et al studied the kinetics of IgM, IgA and IgG responses by an ELISA based on the SARS-CoV-2 core on 208 plasma from 82 confirmed cases and 58 probable cases of COVID-19. The antibodies are found from the first day after the onset of symptoms. The median time to detection of IgM and IgA was 5 days (IQR, 3-6), while IgG was detected 14 days (IQR, 10-18) after onset of symptoms, with a positive rate of 85, 4%, 92.7% and 77.9%, respectively. In confirmed and probable cases, the positive IgM antibody levels were 75.6% and 93.1%, respectively. The detection efficiency by IgM ELISA is superior to that of PCR after 5.5 days of onset of symptoms. The infection detection rate is increased (98.6%) by combining ELISA IgM test with PCR for each patient compared to a single qPCR test (51.9%). No cross-reactivity was found with common coronaviruses.

Zhao et al looked for total antibodies, IgM and IgG in 173 patients (median age, 48 years) with COVID-19 confirmed by PCR. The overall seroconversion rate, IgM and IgG, were 93%, 82.7% and 64.7%, respectively, with a median time to seroconversion around day 12. The presence of antibodies is less than 40% during the week following the onset of the disease to reach 100% (Ab), 94% (IgM) and 80% (IgG) by day 15.

In a study of 285 patients with COVID-19, 100% of patients developed specific antibodies within an average of 19 days after the onset of symptoms. The IgG and IgM antibody plateau is reached six days after seroconversion.

Few data exist on the intra-family spread of the COVID 19 disease, in particular in its minor or moderate form followed on an outpatient basis.

A study, carried out in China, evaluated 318 clusters of at least 3 grouped cases> 3 cases which concerned a total of 1245 cases, occurring in 320 municipalities. The majority of cases are grouped at home (80%) then in transport (26%). Most cases grouped at home concern 3 to 5 cases. Sharing a home appears to be a major risk of contamination.

In Shenzhen, the investigation of 39 COVID / PCR cases and their 1,286 contacts shows a transmission rate (measured by PCR) of 111.2% [9.1 - 13.8]. Transmission rates are important when contacts live in the household or have traveled with the index case.

In France, few data are still available. An epidemiological study, carried out at the end of March 2020, tested 661 people in serology in connection with the high school of Crépy-en-Valois (Oise) where a teacher worked, the first case of French COVID. It appears that the infection attack rate was highest among secondary school staff, teachers and students, and much lower among parents and siblings of students.

The suddenness of the COVID-19 epidemic, its spread, its new character have taken many health care systems to fail.

In the absence of effective treatment against COVID-19 to date, only preventive measures can be effective.

The rapidly epidemic nature and the lack of sufficient protective equipment made it impossible to have perfectly adequate protective measures, even after confinement.

Likewise, in the entourage of a patient with COVID-19, the scarcity of direct diagnostic tests (PCR) from February to April made it possible to diagnose only symptomatic people having recourse to the hospital system or working in a system of care.

For an appropriate public health response, an estimate of the number of people who have encountered the virus and potentially protected is fundamental.

There is little data on exposure to the virus, measured by the presence of specific antibodies in the family circle of an index case.

Several confinement situations in enclosed spaces (cruise ships) have led to transmission rates of around 20%.

The FAMI-CoV study proposes to assess the rate of exposure to the virus in contacts sharing the same focus of index cases. A sub-study will assess the proportion of antibodies that have been neutralizing.

This is a cross-sectional, single-center study carried out on the cohort of index patients followed on an outpatient basis

Recruitment will be done from the active file of patients included in the COVID / PSL cohort or patients followed in city medicine.

Screening This visit makes it possible to offer the study to each patient (INDEX case) corresponding to the inclusion criteria and to their contacts living in the same household on the data recorded in the clinical follow-up files.

It takes place after checking the inclusion and exclusion criteria of subjects. This visit can be done over the phone. The patient information and consent form is issued to the patient or his family.

Inclusion visit and serological test

This visit allows you to:

1. explain the objectives of the study and the test methods
2. give consent and obtain signatures
3. complete the questionnaire for index cases and contacts
4. perform a rapid test looking for anti SARS-CoV-2 antibodies, at the fingertip (sample taken by a professional authorized to perform these tests)
5. reading of the result is immediate
6. the result is given and commented on to each member of the household; they will be kept.

This process is repeated for each index case and each contact case.

Performing the anti-SARS-CoV-2 rapid antibody test Choice of test The COVID-19 IgG / IgM rapid test (whole blood / serum / plasma) (COVID-PRESTO manufactured by the firm AAZ) is a solid phase immunochromatographic test for the rapid, qualitative and differential detection of IgG and IgM antibodies directed against SARSCoV -2 which allows to affirm, in the absence of symptoms, contact with the virus and an acquired immunity a prioriprotective. The test uses anti human IgM antibodies (IgM test line), anti human IgG antibodies (IgG test line) and rabbit IgG (control line (C)) immobilized on a nitrocellulose strip. The conjugate (recombinant COVID-19 antigens labeled with colloidal gold) is also integrated into the strip.

This test was evaluated by 3 laboratories (Bichat Hospital virology laboratory, Orléans laboratory, CNR Lyon reference laboratory Pr B. Lina.

Practice of the test

* The rapid test is performed using a drop of blood obtained at the fingertip (10 microliters) using a lancet.
* The dropper pipette, held vertically, collects the drop of whole blood up to the "sample line"
* Place 1 drop of whole blood (10 μL in the sample well (S) of the cassette.
* Immediately add 2 drops (80μL) of buffer to the well (B) of the cassette.
* Avoid air bubbles; if there is an air bubble, add a 3rd drop of buffer.

The reading is taken after 10 minutes at most by the healthcare professional under medical supervision. Positivity can appear after 1 to 3 minutes.

The reading should not exceed 30 minutes. The rapid tests will be carried out either by authorized personnel who practice them regularly in the context of HIV / Hepatitis screening actions.

In case of sepositivity of the rapid test, it may be offered to index cases and adult contacts, a blood sample of 5 ml of blood for a serothèque allowing a characterization of the antibodies and in particular of the neutralizing antibodies.

ELIGIBILITY:
Inclusion Criteria:

Index case

* Adult> 18 years old
* Having presented a SARS-CoV-2 infection confirmed by PCR (INDEX COVID / PCR +)
* or having presented clinical symptoms compatible with the diagnosis of COVID-19 (COVID-like) with at least 3 of the following symptoms for ⩾ 48 hours: fever, cough, anosmia, ageusia, headache, diarrhea, or CT scan with pneumopathy image in frosted glass
* Living at the time of symptoms with at least 2 other people in the same household
* Written consent for himself and for minors for whom he is responsible

Contact case

* Adult (s) or child (ren), aged 3 to 17 (school age including kindergarten), living in the same household as the index case at the time of the symptoms of the index case
* Written consent for adults
* Consent given by parents for minors

Exclusion Criteria:

* Patient protected by law (patient under guardianship and guardianship, person deprived of liberty)
* Patient with major cognitive disorders.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Measure of the proportion of contact persons who have developed anti-SARS-CoV-2 antibodies (secondary transmission rate) within the same household of a subject who had a COVID-19 disease assessed by a rapid diagnostic-oriented test | 4 hours
  Measure of anti-SARS-CoV-2 antibodies using COVID-PRESTO (AAZ company)

CONTACTS AND LOCATIONS:
Locations (1):
- Christine KATLAMA, Paris, Île-de-France Region, France